CLINICAL TRIAL: NCT01039883
Title: A Phase 1, Randomized, Open-Label, Crossover Safety and Pharmacokinetic Study of 400 mg Albaconazole as a Tablet Formulation Versus a Capsule Formulation in Healthy Subjects
Brief Title: A Study to Compare the Blood Levels of Albaconazole in Healthy Subjects Who Have Received a Single Dose of 400 mg Albaconazole as a Tablet Versus Albaconazole as a Capsule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 114563
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Onychomycosis
Keywords: Healthy Volunteers
MeSH Terms: conditions — Onychomycosis | interventions — albaconazole; Capsules; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Subjects randomized to study product sequence 1 will receive the single albaconazole 400-mg tablet during the first dosing period and the four 100-mg albaconazole capsules during the second dosing period.
  Interventions: Drug: Albaconazole tablet 400mg
- 2 (Experimental): Subjects randomized to study product sequence 2 will receive the four 100-mg albaconazole capsules during the first dosing period and the single albaconazole 400-mg tablet during the second dosing period.
  Interventions: Drug: Albaconazole 100mg capsules, then albaconazole 400mg tablet

INTERVENTIONS:
Drug: Albaconazole tablet 400mg — Albaconazole tablet 400mg single dose, then four albaconazole capsule 100mg single dose
  Other Names: Albaconazole
  Arms: 1
Drug: Albaconazole 100mg capsules, then albaconazole 400mg tablet — Four albaconazole capsule 100mg single dose, then albaconazole tablet 400mg single dose
  Other Names: Albaconazole
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether albaconazole tablets and albaconazole capsules (single 400mg dose) act in the body in the same way over a period of time.

DETAILED DESCRIPTION:
The aim of this study is to compare the bioavailability of the formulation used in earlier clinical studies (albaconazole capsules) with the formulation intended for use in further development (albaconazole tablets). The study is also designed to assess the safety and tolerability of a single oral dose of albaconazole tablets (400 mg), and assess the bioequivalence of albaconazole tablets with albaconazole capsules.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding and willing to provide signed and dated written voluntary informed consent (and any local or national authorization requirements) before any protocol specific procedures are performed.
* Male or female aged from 18 to 45 years at time of consent and at time of first dose.
* A body mass index (BMI) between 18.5 and 30 kg/m2.
* Able to complete the study and to comply with study instructions.
* Free of clinically significant disease as determined by history, physical examination, and laboratory testing.
* The subject is a non-smoker or ex-smoker. If a subject is an ex smoker, he/she must not have used nicotine for at least 6 months before first dose.
* The screening and baseline laboratory parameters must be within normal ranges unless agreed as not clinically relevant by the principal investigator and the sponsor. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, and total bilirubin values should be lower than 1.5 times the upper normal limit at screening.
* The subject will have negative results for the following tests at screening:

  * Hepatitis B surface antigen (HBsAg)
  * Hepatitis B core antibodies (HBcAc)
  * Anti-hepatitis C virus (Anti-HCV)
  * Human immunodeficiency virus (HIV) antibody test
  * Urine drug screen
* Sexually active females of childbearing potential participating in the study must agree to use a medically acceptable method of contraception while receiving protocol-assigned product and until 30 days following the last dose of the study product. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant; including perimenopausal women who are less than 2 years from their last menses. Acceptable contraceptive methods include the following:

  * Hormonal contraception, including oral, injectable, or implantable methods started at least 2 months prior to screening. If hormonal contraception was started less than 2 months prior to screening, then a form of nonhormonal contraception should be added until the third continuous month of hormonal contraception has been completed.
  * Two forms of reliable nonhormonal contraception, to include the use of either an intrauterine device plus a reliable barrier method or 2 reliable barrier methods. Reliable barrier methods include condoms or diaphragms. A cervical cap is also a reliable barrier method, provided that the female subject has never given birth naturally. The combined use of a condom and spermicide constitute 2 forms of acceptable nonhormonal contraception, provided that they are both used properly. The use of spermicide alone and the improper use of condoms are inferior methods of contraception. Subjects with surgical sterilization, including tubal sterilization or partner's vasectomy, must use a form of nonhormonal contraception. A barrier method or sterilization plus spermatocide are acceptable.
* Women who are not currently sexually active must agree to use a medically accepted method of contraception should they become sexually active while participating in the study. Male subjects and/or their partners must use a medically acceptable form of contraception

Exclusion Criteria:

* Female who is pregnant (positive pregnancy test), trying to become pregnant, or breast feeding.
* Received any investigational drug within 30 days of study day 1 or who are scheduled to receive an investigational drug other than the study product during the study.
* Used prescription drug therapy, over the counter (nonprescription) medications, recreational drugs, or herbal products within 30 days of dosing, unless agreed as not clinically relevant by the principal investigator and sponsor.
* Participated in a previous study of the same study product.
* Currently using any medication that, in the opinion of the investigator, may affect the evaluation of the study product or place the subject at undue risk.
* Currently suffering from any disease or condition that, in the opinion of the investigator, may affect the evaluation of the study product or place the subject at undue risk.
* Has a history of anemia, iron deficiency, or iron depletion.
* Has a history of any condition possibly affecting absorption of drug (eg, peptic ulcer disease, gastrectomy, intestinal malabsorption).
* Considered immunocompromised.
* History of drug, prescription medicine, or alcohol abuse within the past 2 years.
* Has a history of known or suspected intolerance to any of the ingredients of the study products.
* Has known drug allergies.
* Has a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, or connective tissue diseases or disorders.
* Intends to donate blood or blood components while receiving the study product or for the duration of the pharmacokinetic sampling period.
* Has donated blood or has had significant blood loss (≥250 mL) within 30 days before dosing or has donated plasma within 7 days before dosing.
* Has QT interval corrected for heart rate (Fridericia's correction formula) (QTcF) >450 ms or any ECG abnormality except for the following:

  * Mild sinus bradycardia in younger, athletic subjects (heart rate down to 46 beats per minute allowed).
  * Mild sinus arrhythmia.
  * Mild first degree atrioventricular (A-V) block (P-R interval <0.23 sec).
  * Mild right or left axis deviation.
  * Incomplete right bundle branch block.
  * Isolated left anterior fascicular block (left anterior hemiblock) in younger, athletic subjects.
  * Early repolarization.
  * Uncorrected QT interval or QT interval corrected for heart rate with Bazett's correction formula (QTcB) exceeding 450 ms, with a QTcF ≤450 ms.
* Considered unable or unlikely to attend the necessary visits.
* Employees of investigator/ clinical research organization or Stiefel involved in the study, or an immediate family member (partner, offspring, parents, siblings, or sibling's offspring) of an employee involved in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-11-23 (Actual); Primary Completion 2010-01-20 (Actual); Study Completion 2010-01-20 (Actual)

PRIMARY OUTCOMES:
Bioavailability of albaconazole | Blood samples taken predose and at 30 minutes, and 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12 (day 1 time points), 18 (day 2), 24 (day 2), hours post-dose and once a day on days 3-16

SECONDARY OUTCOMES:
Safety and tolerability of a single oral dose of 400mg albaconazole tablet | ECGs and lab tests at screening, pre-dose, and 3 hours, and 16 days post-dose. Physical examination at screening, pre-dose and 16 days post-dose. Assessment of adverse events from consent to 16 days post-dose (second dosing period).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Buffalo Clinical Research Center, Buffalo, New York, United States

REFERENCES:
- [Background] van Rossem K, Lowe JA. A Phase 1, randomized, open-label crossover study to evaluate the safety and pharmacokinetics of 400 mg albaconazole administered to healthy participants as a tablet formulation versus a capsule formulation. Clin Pharmacol. 2013;5:23-31. doi: 10.2147/CPAA.S39600. Epub 2013 Jan 30. PMID 23390369
- See also: Results for study 114563 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114563?search=study&study_ids=114563#rs